CLINICAL TRIAL: NCT00223496
Title: 12- Week Open Label Treatment of Refractory Bipolar Depression (BD) With Combination of Depakote ER (DEP) and Aripiprazole (AZP)
Brief Title: 12- Week Open Label Treatment of Refractory Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Charles L. Bowden, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0340013419
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Depression; Refractory
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aripiprazole (Experimental): Aripiprazole open-label in doses ranging from 5-30mg QD adjunct to Divalproex 500-2500mg QD.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole5mg - 30mg, every day (QD), for 12 weeks.

SUMMARY:
1. Determine the change in symptomatology and function in refractory bipolar depression, when treated with combination of DEP+AZP for a period of 12 weeks
2. Determine the tolerability and safety of AZP added to DEP in the treatment of refractory bipolar depression

DETAILED DESCRIPTION:
)Determine the change in symptomatology and function in refractory bipolar depression, when treated with combination of DEP+AZP for a period of 12 weeks

2) Determine the tolerability and safety of AZP added to DEP in the treatment of refractory bipolar depression

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar disorder I or II according to M.I.N.I.
* patient has signed informed consent
* male, or female who is using effective birth control if of child bearing age
* age 18 and above
* currently in a depressed phase, with or without psychotic features, of the illness based on DSM-IV/MINI criteria
* score of more than 19 on the MADRS
* history of treatment refractory bipolar depression as defined by failure of the depressive episode to respond to a mood stabilizer alone or a combination of 2 or more mood stabilizers or a combination of a mood stabilizer and an antidepressant

Exclusion Criteria:

* current liver disease,
* illness precluding the use of depakote er
* patients who have been treated with a DEP and AZP combination in the past
* Alcohol/drug dependence in the past one month
* CNS neoplasms, demyelinating diseases, degenerative neurological condition or active CNS infection
* history of seizure, known EEG with frank paroxysmal activity, known CT of brain showing gross structural abnormalities, cerebral vascular disease by history or structural brain damage from trauma
* thyroid dysfunction
* unstable general medical condition
* require antipsychotic other than abilify

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Singh, MD, Principal Investigator — University of Texas; Charles L Bowden, MD, Principal Investigator — University of Texas
Locations (1):
- Univ of Texas Helath Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from March 2006 to June 2009 from clinic patients and those responding to public advertisements.
Pre-assignment Details: Subjects who entered study in a bipolar depressed state were started on divalproex ER. Those still depressed, according to depression rating scales, after visit 4 were given aripiprazole in addition to divalproex ER.
Groups:
- Aripiprazole Plus Divalproex ER: Study recruited subjects with bipolar disorder who were currently in a depressed state according to rating scales. Subjects were started on divalproex. After 3 weeks on divalproex if patients were still exhibiting depression symptoms then they were started on aripriprazole in addition to divalproex. Those subject who were no longer in a depressed state were terminated from study. Subjects proceeded in study on both medications and were assessed by physician for depression and mania symtpoms using rating scales, until end of study.
Period: Overall Study
Arm/Group | Aripiprazole Plus Divalproex ER
Started | 32 (32 people consented, 19 were baselined)
Completed | 10
Not Completed | 22
Not completed — screen failure | 9
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: 32 subjects consented, 19 subjects were baselined
Groups:
- Aripiprazole: Study recruited subjects with bipolar disorder who were currently in a depressed state according to rating scales. Subjects were started on divalproex. After 3 weeks on divalproex if patients were still exhibiting depression symptoms then they were started on aripriprazole in addition to divalproex. Those subject who were no longer in a depressed state were terminated from study. Subjects proceeded in study on both medications and were assessed by physician for depression and mania symtpoms using rating scales, until end of study.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Primary Measure:Reduction in Depression Symptoms
Description: Primary efficacy will be assessed by the proportion of patients achieving a 50% reduction (range 0- 60, higher the number the more depressed) on the Montgomery Asberg Depression Rating Scale (MADRS) (defined as response) concomitant with a Clinical Global Impression Scale(CGI-S) improvement of 1 or 2 (range 0-7, higher the number the more severe the overall bipolar symptoms).
Time Frame: up to 12 weeks
Measure: Number; unit: participants
Groups:
- Aripiprazole Plus Divalalproex ER: Study recruited subjects with bipolar disorder who were currently in a depressed state according to rating scales. Subjects were started on divalproex. After 3 weeks on divalproex if patients were still exhibiting depression symptoms then they were started on aripriprazole in addition to divalproex. Those subject who were no longer in a depressed state were terminated from study. Subjects proceeded in study on both medications and were assessed by physician for depression and mania symtpoms using rating scales, until end of study.
Arm/Group | Aripiprazole Plus Divalalproex ER
Number analyzed (Participants) | 16
participants | 16

ADVERSE EVENTS:
Time Frame: 3-31-2006 to 9-11-2009, 3 yrs 6 mo
Description: Patient reporting and systematic questioning
Arm/Group | Aripiprazole Plus Divalproex ER
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Plus Divalproex ER (N=16)
Akathisia (Nervous system disorders) | 6 (6) — a feeling of restlessness that results in movements of body parts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No